CLINICAL TRIAL: NCT04214743
Title: Ocular Microvascular Changes in Patients With Sepsis
Status: Completed | Type: Observational
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Research Council of Lithuania (Other)
Responsible Party: Principal Investigator, Andrius Pranskunas, MD, Lithuanian University of Health Sciences
Other Study IDs: 2018/BE-2-18
Record Dates: First submitted 2019-12-28; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Sepsis; Retinal Microcirculation Disorder; Conjunctiva; Disorder
Keywords: Conjunctival microcirculation; retinal vessels; fundus imaging; IDF imaging; sepsis
MeSH Terms: conditions — Sepsis; Conjunctival Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Incident dark field videomicroscope from Braedius — It allows to look at conjunctival microcirculation
Device: Fundus camera from Optomed — It allows to monitor retinal microvasculature

SUMMARY:
This study evaluates differences in the ocular microcirculation between septic patients and healthy subjects and the course of ocular microvasculature in survivors and non-survivors over a 24 hours period of time in septic patients

DETAILED DESCRIPTION:
Conjunctival imaging, using IDF video microscope, and retinal imaging, using portable digital fundus camera, as well as systemic hemodynamic measurements, were performed in septic patients at three time points: at baseline, 6 hours and 24 hours. Baseline conjunctival and retinal microcirculatory parameters were compared with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with sepsis or septic shock within the first 24 hours after ICU admission

Exclusion Criteria:

* psychiatric disorders, brain diseases, chronic alcoholism, autoimmune rheumatic diseases
* ophthalmological diseases, such as glaucoma, age-related macular degeneration, diabetic retinopathy and cataract

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with sepsis or septic shock within the first 24 hours after ICU admission
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Microvascular flow index in conjunctival small vessels | 24 hours
  Differences in MFI in conjunctival small vessels between septic patients and healthy controls and differences between survivors and non-survivors

SECONDARY OUTCOMES:
Central retinal arteriolar equivalent of retinal vessels | 24 hours
  Differences in central retinal arteriolar equivalent of retinal vessels between septic patients and healthy controls and differences between survivors and non-survivors

CONTACTS AND LOCATIONS:
Overall Officials: Andrius o Pranskunas, Principal Investigator — Lithuanian University of Health Sciences
Locations (1):
- Hospital of Lithuanian university of health sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simkiene J, Pranskuniene Z, Vitkauskiene A, Pilvinis V, Boerma EC, Pranskunas A. Ocular microvascular changes in patients with sepsis: a prospective observational study. Ann Intensive Care. 2020 Apr 7;10(1):38. doi: 10.1186/s13613-020-00655-x. PMID 32266602